CLINICAL TRIAL: NCT05368116
Title: Effectiveness of Video Assisted Self Management Program on Chemotherapy Side Effects in Terms of Knowledge, Self Efficacy and Severity of Side Effects Among the Cancer Patient Receiving Chemotherapy at Oncology Day Care
Brief Title: Effectiveness of Video Assisted Self Management Program on Chemotherapy Related Side Effects .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ILBS-VASMPCa-103
Record Dates: First submitted 2022-05-09; First posted 2022-05-10 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-03

CONDITIONS: Cancer Patients
Keywords: Video Assisted Self Management Program; Knowledge; Self Efficacy; Cancer Patients; Chemotherapy; Severity
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Assisted Self Management Program (Experimental): It is the systematically designed Video Assisted teaching program to educate cancer patients receiving chemotherapy under the experimental group about the management of chemotherapy related side effects at home .It will be one to one teaching session of 10-20 minutes conducted by the principal researcher with the help of a video on self management of chemotherapy related side effects and the video will focus on the self management of selected side effects of chemotherapy including Nausea, vomiting, Diarrhea, Constipation, Fever, Mucositis, Skin changes, and Alopecia related distress.
  Interventions: Other: Video Assisted Self Management Program
- Standard of Care (Active Comparator): The participants were given video when they come to oncology day care and instruct the participants to watch the video at home. Knowledge, self efficacy and severity of chemotherapy related side effects were assessed after one week.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Video Assisted Self Management Program — The main aim of this intervention is to educate the cancer patients receiving chemotherapy regarding the management of chemotherapy related side effects.
  It will be one to one teaching session of 10-20 minutes conducted by the principal researcher with the help of a video on self management of chemotherapy related side effects and the video will focus on the self management of selected side effects of chemotherapy including nausea vomiting , Diarrhea , Fever , Mucositis , Skin changes , and Alopecia related distress.
  The participants were given video when they comes to the Oncology day care and researcher instructs the participants to watch the video and at the same time the doubts asked by the participants were cleared by the researcher.
  Arms: Video Assisted Self Management Program
Other: Standard of care — Standard of care
  Arms: Standard of Care

SUMMARY:
A study to assess the effectiveness of video assisted Self Management Program on chemotherapy side effects in terms of Knowledge, Self Efficacy and Severity of side effects among the Cancer patient receiving chemotherapy at Oncology day care ILBS , New Delhi.

Primary Objective:

1. To assess the Knowledge, Self Efficacy and Severity of side effects of chemotherapy related side effects in the Experiment Vs. Comparison group among the cancer patients receiving chemotherapy.
2. To compare the knowledge and self efficacy scores in Experimental Vs. Comparison group after video assisted SMP among the cancer patients receiving chemotherapy.
3. To compare the severity of chemotherapy related side effects in Experiment Vs. Comparison group before and after video assisted SMP among the cancer patients receiving chemotherapy.

Secondary Objective To find the correlation between knowledge and self efficacy scores among the cancer patients receiving chemotherapy under Experimental Group.

2. To determine the association of Severity of side effects with the knowledge and self efficacy scores among the cancer patients receiving chemotherapy.

3. To determine the association of knowledge, self efficacy with the socio demographic and clinical variables among the cancer patients receiving chemotherapy.

The study assumes that:

1. Video assisted teaching is an accepted teaching strategy and enhances teaching learning activities.
2. Patients may have limited knowledge about the management of side effects related to chemotherapy including nausea, vomiting, diarrhea, Constipation, dry skin, fever, alopecia related distress and pain.
3. Patients may have decrease severity of chemotherapy related side effects including nausea, vomiting, diarrhea, Constipation , dry skin, fever , alopecia related distress and pain. After the self management program.

DETAILED DESCRIPTION:
Effectiveness A measure of the extent to which a specific intervention, procedure, regimen, or service when deployed in the field of routine circumstances, does it intended to do for a specific population. (Wojtezak, 2002) In this study, effectiveness refers to the degree to which the video assisted SMP is successful in the management of chemotherapy related side effects in terms of gain in Knowledge, self efficacy scores and reducing the severity of side effects among the cancer patient receiving chemotherapy.

Video Assisted Self Management Program It referred to an instructional aid which incorporates visual and auditory information on a topic for individual to understand and learn. (MedCrave 2016) In this study it refers to the systematically designed Video Assisted teaching program to educate cancer patients receiving chemotherapy under the experimental group about the management of chemotherapy related side effects at home .It will be one to one teaching session of 10-20 minutes conducted by the principal researcher with the help of a video on self management of chemotherapy related side effects and the video will focus on the self management of selected side effects of chemotherapy including Nausea, vomiting , Diarrhea ,Constipation, Fever , Mucositis , Skin changes , and Alopecia related distress.

Chemotherapy side effects It is the unintended effect occurring at normal dose related to the pharmacological properties. (WHO) In this study it refers to the commonly reported chemotherapy related side effects by the patients receiving chemotherapy including nausea vomiting, Diarrhea, Constipation, Fever, Mucositis, Dry skin, and Alopecia related distress in cancer patients after receiving chemotherapy.

Knowledge It is defined as the familiarity, awareness, or understanding of someone or something such as facts, skills or objects. (Plato) In this study it refers to the correct response of the patient to the questionnaire regarding the self management of the side effects of chemotherapy. It will be assessed by the Structured Questionnaire on self management of chemotherapy related side effects with 20 items. The scores will be analyzed in the form of means.

Cancer Patients Cancer Patient is defined as a person receiving or registered to receive medical treatment in the Hospital for Cancer. (American Cancer Society) In this study it refers to the person either male or female who is suffering from any type of cancer that includes but not limited to Head and Neck, Pancreas, Liver, Gall bladder, Breast, Stomach, and mouth cancer and receiving chemotherapy at Onco day care ILBS, New Delhi at the time of data collection.

Self Efficacy It refers to an individual's belief in his or her capacity to execute behaviors necessary to produce specific performance attainments. It reflects confidence in the ability to exert control over one's own motivation, behavior and social environment. (Bandura, 1977) In this study it refers to the level of confidence of the cancer patients about their ability to manage the chemotherapy related side effects at home. It will be assessed by the structured symptom management self efficacy tool consisting of Twelve items. The mean score of self efficacy will be used to compare the Experimental and Comparison groups.

Severity of Chemotherapy Related Side Effects It refers to the degree to which a single side effect affects the patient graded on a scale of three. (Aakshdeep batra AIIMS) In this study it refers to the magnitude or the intensity (Grading) of the chemotherapy related side effects among the cancer patients receiving chemotherapy. It will be assessed by the Common Terminology Criteria for the Adverse Events (CTCAE) Version -5 and the Chemotherapy related side effects will be assessed in terms of their presence and the severity from the day of last chemotherapy cycle to the day of present cycle. It will be a recall basis assessment.

Hypothesis

All hypotheses were tested at 0.05 level of significance:

H1: There will be a significant difference between the Experimental and comparison group in terms of their mean gain in knowledge scores after video assisted SMP as assessed by the structured knowledge questionnaire.

H2 : There will be a significant difference between the Experimental and Comparison group in terms of their mean gain in Self efficacy scores after video assisted SMP as assessed by the self efficacy scale.

H3: There will be a significant difference between the Experimental and Comparison group in terms of their mean scores of Severity of the side effects after video assisted SMP as assessed by the CTCAE criteria.

H4: There will be a significant correlation of knowledge and self Efficacy scores in Experimental group among the cancer patients receiving chemotherapy.

H5: There will be a significant association of severity of chemotherapy related side effects with the knowledge and self efficacy scores among the cancer patients receiving chemotherapy.

H6: There will be a significant association of knowledge and self efficacy scores with the sociodemographic and clinical variables among the cancer patients receiving chemotherapy.

Delimitations of the study The study was delimited to

• Patients who are receiving chemotherapy at Oncology Day care in ILBS, New Delhi.

Variables under Study Independent Variables In the present study, the independent variable was the Video assisted Self Management Program. The protocol used in this study was prepared after an extensive review of literature.

Dependent Variables In the present study, the dependent variables were Knowledge, self efficacy and severity.

Socio Demographic Variables In the present study, the socio demographic variables studied were Age, Gender, Marital status, Education, Occupation, Religion, Family monthly income.

Clinical Variables The clinical variables are Type of Cancer, duration of time since diagnosis, Last chemotherapy cycle received, Stage of cancer , No of present chemotherapy cycle received, Any Family members/ closed relatives / friends received chemotherapy ever , Any training received on management of side effects.

Research Settings The setting for the present study is Institute of Liver and Biliary Sciences. It is a super specialty hospital specialized in Liver and biliary sciences .The hospital has facilities like Emergency Unit, Transplant Intensive care Unit, Operation Theatres, Liver coma Intensive care Unit. The hospital also has the facility of Onco Day care where chemotherapy is provided.

The study was conducted at the Oncology Day care. The Oncology Day care unit is a 9 bedded unit. The rationale for selecting the setting was easy availability of the sample of interest , feasibility of conducting the study and familiarity with the setting.

Intervention Description of Video Assisted Self Management Program It is a intervention which was designed by the principal investigator In this study it refers to the systematically designed Video Assisted teaching program to educate cancer patients receiving chemotherapy under the experimental group about the management of chemotherapy related side effects at home. After extensive review of literature under the guidance of guide and Medical Oncologist. The Video Assisted teaching program was validated by the Medical oncologist and other experts.

The main aim of this intervention is to educate the cancer patients receiving chemotherapy regarding the management of chemotherapy related side effects.

It will be one to one teaching session of 10-20 minutes conducted by the principal researcher with the help of a video on self management of chemotherapy related side effects and the video will focus on the self management of selected side effects of chemotherapy including nausea vomiting , Diarrhea , Fever , Mucositis , Skin changes , and Alopecia related distress.

The participants were given video when they comes to the Oncology day care and researcher instructs the participants to watch the video and at the same time the doubts asked by the participants were cleared by the researcher.

ELIGIBILITY:
Inclusion Criteria:

All the cancer patients receiving chemotherapy at Onco day care ILBS which will be included in the study who-

* Were 18 years or older
* Patients who have undergone at least one chemotherapy cycle.
* Patients who are stable.
* Can Communicate in English / Hindi
* Patients who are Mentally alert

Exclusion Criteria:

All cancer patients undergoing chemotherapy was excluded from the study who -

* Patients who are Android mobile users Patients with visual and hearing impairments
* Had hemodynamic instability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Knowledge regarding the management of chemotherapy related side effects. | up to 5 weeks
  A structured 20 item knowledge questionnaire developed for assessment of knowledge among the cancer patients receiving chemotherapy at Onco day care Ilbs. The knowledge questionnaire will be self reported by the subjects.
self efficacy in relation to symptom management relevant to chemotherapy for patients with cancer. | up to 5 weeks
  The Structured Symptom-Management Self-Efficacy Scale derived from - Symptom-Management Self-Efficacy Scale Breast Cancer (SMSES-Breast Ca.) It was developed by SY Liang et al., in 2015 that measure perceived self efficacy in terms of respondent's ability to self manage the symptoms of chemotherapy. It is an 11-point Likert scale was used for each item that ranged from 0 (not confident at all) to 10 (completely confident), with higher scores representing higher perceived self-efficacy.
Severity of Side effects including Nausea, Vomiting, Diarrhea, Constipation, Mucositis, Fever, Pain ,Dry Skin and alopecia related distress. | up to 5 weeks
  It consists of grades which are used to assess the severity of adverse events. Grades ranges from 0 to 5. The scores assessed by the researcher for the severity of side effects will be verified by the doctors on duty.
  The Distress thermometer was developed as a simple tool to effectively screen for symptom of Alopecia related distress. It is a self reported tool using a 0-10 rating scale. The scale was explained to all the participants and participants were asked to circle or pick a number 0-10 from the drop down box that best describes how much distress patient have been experiencing in the past weeks including today.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Ms Bisht, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India